CLINICAL TRIAL: NCT05753904
Title: The Impact of Conjoint Tendon Resection on Functional Internal Rotation of the Shoulder Following Reverse Shoulder Arthroplasty: A Prospective, Randomized Clinical Trial
Brief Title: Conjoint Tendon Resection During Reverse Total Shoulder Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator No Longer at Institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2094589
Record Dates: First submitted 2023-02-12; First posted 2023-03-03 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Injuries; Patient Satisfaction; Internal Rotation Contracture-shoulder
Keywords: Reverse Total Shoulder Arthroplasty; Functional Internal Rotation; Conjoint Tendon
MeSH Terms: conditions — Shoulder Injuries; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized-controlled clinical trial comparing standard of care RTSA to RTSA with conjoint tendon resection in 64 patients undergoing RTSA by a single surgeon.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors will not be blinded to intervention. The primary outcome is postoperative functional internal rotation. Secondary outcome measures include VAS, ASES, SANE, PROMIS, and VR-12 scores, as well as forward elevation and external rotation at the side, and complications at any time point. Our null hypothesis is that patients who undergo conjoint tendon resection during RTSA will have significantly increased functional internal rotation and clinically significant improved above-mentioned scores compared to non-resected tendon patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse Total Shoulder Arthroplasty (No Intervention): For RTSA using a deltopectoral approach, the Perform glenoid and humeral components of Tornier Stryker Reverse Shoulder system will be used for all cases. The sizes and offsets of the components will be chosen based on each patient's local anatomy which will vary among patients. The subscapularis tendon will be repaired using three transosseous nonabsorbable sutures whenever there is a reparable subscapularis tendon. After definitive implantation of the prosthesis is completed, in the 'no interventional' group, the wound will be closed in layers, and the shoulder will be immobilized in an abduction sling.
- Reverse Total Shoulder Arthroplasty with Conjoint Tendon Resection (Experimental): RTSA in the experimental group will be identical, except for that after definitive implantation of the prosthesis is completed, in the 'experimental' group, the conjoint tendon will be released completely via a transverse incision made at a level 2 cm distal to the coracoid process for the patients assigned the conjoint resection group. Electrocautery will be used for the resection, and the underlying muscular portion of the conjoint tendon will be preserved. As mentioned above, the control group will not receive this conjoint tendon resection. Similarly, in the experimental group, the wound will be closed in layers, and the shoulder will be immobilized in an abduction sling.
  Interventions: Procedure: Conjoint Tendon Resection

INTERVENTIONS:
Procedure: Conjoint Tendon Resection — For conjoint tendon resection in the experimental group, the conjoint tendon will be released completely via a transverse incision made at a level 2 cm distal to the coracoid process for the patients assigned the conjoint resection group. Electrocautery will be used for the resection, and the underlying muscular portion of the conjoint tendon will be preserved.
  Arms: Reverse Total Shoulder Arthroplasty with Conjoint Tendon Resection

SUMMARY:
Reverse total shoulder arthroplasty (RTSA) can reliably restore active forward elevation, abduction, and external rotation, which are often lost in patients with massive rotator cuff tears. However, functional internal rotation (i.e., functional movements of the hand behind the body) is often unsatisfactorily restored and/or lost after RTSA. This study aims to compare the standard surgical approach for RTSA to RTSA with conjoint tendon resection with the targeted metric being postoperative functional internal rotation.

DETAILED DESCRIPTION:
This study will be a prospective, randomized-controlled clinical trial comparing standard of care RTSA to RTSA with conjoint tendon resection in 64 patients undergoing RTSA by a single surgeon. Participants and assessors will not be blinded to intervention. The primary outcome is postoperative functional internal rotation. Secondary outcome measures include VAS, ASES, SANE, PROMIS, and VR-12 scores, as well as forward elevation and external rotation at the side, and complications at any time point. Our null hypothesis is that patients who undergo conjoint tendon resection during RTSA will have significantly increased functional internal rotation and clinically significant improved above-mentioned scores compared to non-resected tendon patients.

ELIGIBILITY:
Inclusion criteria

- All patients undergoing primary reverse total shoulder arthroplasty (RTSA)

Exclusion criteria

* Revision RTSA
* RTSA for acute proximal humerus fracture or fracture sequela

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data collection for individual participant data will primarily be electronically based and not available to members outside of the research team. A breach of confidentiality and/or privacy is a risk of this study. To prevent this, all collected data will be stored electronically in password-protected files to protect patient identity and information. All information will be collected and reviewed by the research team only. Data will be maintained on a password-protected computer that will be accessible only to the study team. No patient identifiers will be maintained in the database. Every attempt will be made to minimize missing data. Multiple contact details will be taken at recruitment, and a system of reminders plus phone contact if applicable will be made to ensure patients make follow-up appointments.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reverse Total Shoulder Arthroplasty | Reverse Total Shoulder Arthroplasty With Conjoint Tendon Resection
Started | 13 | 13
Completed | 9 | 8
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reverse Total Shoulder Arthroplasty | Reverse Total Shoulder Arthroplasty With Conjoint Tendon Resection | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.46 (6.881785696) | 69.97 (5.241598895) | 70.71 (6.049666234)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Functional Internal Shoulder Rotation
Description: . Functional internal rotation will be measured based on the highest anatomical level that the patient's thumb can reach:
  * Side
  * Ipsilateral buttock
  * Lower lumbar
  * Mid-lumbar
  * Upper lumbar
  * Thoracolumbar junction
  * T10 and above
Time Frame: Functional Internal Shoulder Rotation will be measured at the 6 Month FU
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team.
Measure: Number; unit: participants
Arm/Group | Reverse Total Shoulder Arthroplasty | Reverse Total Shoulder Arthroplasty With Conjoint Tendon Resection
Number analyzed (Participants) | 3 | 4
participants
  Side | 1 | 1
  Ipsilateral buttock | 1 | 2
  Lower Lumbar | 0 | 0
  Mid-Lumbar | 1 | 1
  Upper Thoracic | 0 | 0
  Thoracolumbar | 0 | 0
  T10 and Above | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events among participants
Arm/Group | Reverse Total Shoulder Arthroplasty | Reverse Total Shoulder Arthroplasty With Conjoint Tendon Resection
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT05753904/Prot_SAP_000.pdf